CLINICAL TRIAL: NCT04158349
Title: Phase I Trial of Intraperitoneal Oxaliplatin in Combination With Intravenous mFOLFIRI for Peritoneal Carcinomatosis From Colorectal and Appendiceal Cancer
Brief Title: Intraperitoneal Oxaliplatin in Combo w IV mFOLFIRI for Peritoneal Carcinomatosis From Colorectal & Appendiceal Cancer
Acronym: IPOX-FOLFIRI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Decision
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCI126164
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Appendiceal Cancer; Peritoneal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Appendiceal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multi-center, open-label phase I trial designed to determine the MTD of IP oxaliplatin when given in combination with mFOLFIRI. This will be conducted according to a traditional 3+3 dose-escalation schedule and halted once MTD is established.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 0 (Experimental): Dose Level 0: 85 mg/m2 Oxaliplatin IP every 2 weeks
  Interventions: Drug: Oxaliplatin; Drug: mFOLFIRI
- Dose Level 1 (Experimental): Dose Level 1: 95 mg/m2 Oxaliplatin IP every 2 weeks
  Interventions: Drug: Oxaliplatin; Drug: mFOLFIRI
- Dose Level 2 (Experimental): Dose Level 2: 105 mg/m2 Oxaliplation IP every 2 weeks
  Interventions: Drug: Oxaliplatin; Drug: mFOLFIRI

INTERVENTIONS:
Drug: Oxaliplatin — Subjects will be accrued in cohorts of 3 to 6 subjects per dose level starting at Dose Level 0 (85 mg/m2). Escalation will continue as described in the protocol until DLT stopping rules are met or the highest dose level is reached.
Drug: mFOLFIRI — mFOLFIRI is a standardized chemotherapy regimen utilizing 5-fluorouracil, leucovorin, and irinotecan administered on day one of a 14-day cycle. 5-Fluorouracil, leucovorin, and irinotecan should be prepared and administered per the package insert and local institutional guidelines.

SUMMARY:
This study is a prospective, multi-center, open-label phase I trial designed to determine the maximun tolerated dose of IP oxaliplatin when given in combination with mFOLFIRI.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, open-label phase I trial designed to determine the MTD of IP oxaliplatin when given in combination with mFOLFIRI. This will be conducted according to a traditional 3+3 dose-escalation schedule and halted once MTD is established.

After consent and once deemed eligible for trial participation, patients will receive four cycles of study therapy. During therapy, patients will be monitored for dose-limiting toxicities and adverse events. After completion of all four cycles patients will be followed until resolution of any ongoing study treatment-related adverse events, initiation of alternative treatment, and survival.

Study drug treatment will be administered on day one of a 14-day cycle and the DLT evaluation period will be defined as the first three cycles of combination treatment (from cycle one day one to the last day of cycle three). The severity of AEs will be graded according to the NCI-CTCAE version 5.0 A standard 3+3 dose escalation design will be used to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) while ensuring the safety and tolerability of the treatment. The study will test three dose levels of oxaliplatin.

Dose Level 2 105 mg/m2 IP every 2 weeks Subjects will be accrued in cohorts of 3 to 6 subjects per dose level starting at Dose Level 0 (85 mg/m2). Escalation will continue until DLT stopping rules are met or the highest dose level is reached.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Histopathologically or cytologically confirmed unresectable colon, rectal or appendiceal adenocarcinoma with synchronous or metachronous (defined as occurring > 6 months after initial diagnosis) peritoneal dissemination of disease. (Stage IV peritoneal-based disease only)
* Patient has active, measurable disease as defined by RECIST 1.1 and assessed by either abdominal CT/MRI.
* Patients must be willing and able as assessed the treating investigator to undergo placement of an IP catheter and a Port-A Cath, if not already present.
* Patients must have known satisfactory cardiopulmonary function as assessed by the treating investigator.
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) > 1200/mm3
    * Platelet count > 100,000/mm3
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN
  * Coagulation:

    * International normalized ratio (INR) ≤ 1.5
    * Patients who are therapeutically anticoagulated and whose antithrombotic treatment can be withheld for operation are eligible.
  * Renal:

    * BUN and serum creatinine within normal limits.
    * eGFR ≥50 mL/min/1.73m2 or creatinine clearance ≥50 mL/min by Cockcroft-Gault
* Negative serum or urine pregnancy test at screening for women of childbearing potential.
* Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last study treatment administration if the risk of conception exists.
* Recovery to baseline or ≤ Grade 1 CTCAE v.5 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* Willing to return for follow-up.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

Sensory neuropathy > grade 1 from prior therapy.

* Known low or absent Dipyrimidine Dehydrogenase (DPD) activity.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Patients with metastases outside the peritoneal cavity.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
  * Other clinically significant disorders that would preclude safe study participation.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  -Note: Patients on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Known chronic hepatitis B virus (HBV) or hepatitis C virus infection with a detectable viral load.

  -Note: Patients with an undetectable HBV viral load on appropriate suppressive therapy are eligible. Patients with an undetectable HCV viral load on appropriate treatment are eligible.
* Live vaccinations, except flu and COVID within 4 weeks of cycle one day one and while on trial.
* Known prior severe hypersensitivity to platinum compounds, any of the investigational medication or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.4.2. A washout period of prohibited medications for a period of at least 5 half-lives or 4 weeks, whichever is shorter, should occur prior to the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Assess the maximum tolerated dose of intraperitoneal (IP) oxaliplatin with systemic IV 5-fluorouracil, leucovorin, and irinotecan (mFOLFIRI) every 2 weeks in patients with unresectable peritoneal carcinomatosis of colorectal or appendiceal origin | One Cycle is 14 days. The DLT evaluation period will be defined as the first three cycles of combination treatment (from cycle one day one to the last day of cycle three (42days)
  The incidence of DLTs during the defined DLT period

SECONDARY OUTCOMES:
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment and the IP catheter will be measured. | up to 3 years
  To assess the safety and feasibility of IP oxaliplatin when administered with systemic mFOLFIRI in patients with peritoneal carcinomatosis of colorectal or appendiceal origin.
The efficacy of IP oxaliplatin plus systemic mFOLFIRI in patients with peritoneal carcinomatosis of colorectal or appendiceal origin will be measured. | up to 3 years
  • Objective response rate (ORR) after four cycles of study therapy. ORR will be assessed by the number of patients obtaining a complete response plus the number of patients obtaining a partial response divided by the number of total response evaluable subjects.
The efficacy of IP oxaliplatin plus systemic mFOLFIRI in patients with peritoneal carcinomatosis of colorectal or appendiceal origin will be measured. | Up to 3 years
  • Overall survival (OS) will be assessed as the time from trial initiation until death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lambert, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No